CLINICAL TRIAL: NCT00830219
Title: The Relative Bioavailability Study of Two Ropinirole 0.25 mg Tablets Under Fed Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teva Pharmaceuticals USA (Industry)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 10436009
Record Dates: First submitted 2009-01-26; First posted 2009-01-27 (Estimated); Results first posted 2009-08-18 (Estimated); Last update posted 2009-09-15 (Estimated); Status verified 2009-09

CONDITIONS: Healthy
Keywords: Bioequivalence; Healthy Subjects
MeSH Terms: interventions — ropinirole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Ropinirole HCl 0.25 mg Tablets
- 2 (Active Comparator)
  Interventions: Drug: Requip® 0.25 mg Tablets

INTERVENTIONS:
Drug: Ropinirole HCl 0.25 mg Tablets — 1 x 0.25 mg, single dose fed
  Arms: 1
Drug: Requip® 0.25 mg Tablets — 1 x 0.25 mg, single dose fed
  Arms: 2

SUMMARY:
The purpose of this study is to compare relative bioavailability of the test formulation of ropinirole hydrochloride 0.25 mg tablets (Manufactured and distributed by TEVA Pharmaceuticals USA) with the already approved formulation REQUIP® (ropinirole hydrochloride) 0.25 mg tablets (GlaxoSmithKline) under fed conditions in healthy, adult subjects.

DETAILED DESCRIPTION:
Criteria for Evaluation: FDA Bioequivalence Criteria

Statistical Methods: FDA bioequivalence statistical methods

ELIGIBILITY:
Inclusion Criteria:

* Males and females, 18 to 45 years of age (inclusive), with a body mass index (BMI) of 19-30 kg/m² inclusive and weighing at least 120 lbs.
* Sitting (at least 5 minutes) blood pressure of at least 100/70 and sitting pulse of at least 60 b.p.m.
* Good health as determined by lack of clinically significant abnormalities in health assessments performed at screening.
* Signed and dated informed consent form, which meets all criteria of current FDA regulations.
* If female and of child bearing potential, subjects must be prepared to abstain from sexual intercourse or use a reliable barrier method of contraception (e.g. condom with spermicide, IUD) during the duration of the study. Female subjects who have used oral contraceptives within 14 days or injected or implanted hormonal contraceptives within 180 days of dosing will not be allowed to participate.

Exclusion Criteria:

* If female, pregnant, lactating, or likely to become pregnant during the study.
* History of allergy or sensitivity to ropinirole or other dopamine agonists (e.g. Corolpam®, Dostinex®, Mirapex®, Permax®, Symmetrel®) or history of any drug hypersensitivity or intolerance which, in the opinion of the investigator, would compromise the safety of the subject or the study.
* History of dizziness, lightheadedness or fainting upon standing.
* Significant history or current evidence of chronic infectious disease, system disorders, organ dysfunction, hyper/hypotension, arrhythmia, tachycardia, seizure disorder or glaucoma.
* Presence of gastrointestinal disease or history of malabsorption within the last year.
* History of psychiatric disorders occurring within the last two years that required hospitalization or medication.
* Presence of a medical condition requiring regular treatment with prescription drugs.
* Use of pharmacologic agents known to significantly induce or inhibit drug metabolizing enzymes within 30 days prior to dosing.
* Receipt of any drug as part of a research study within 30 days prior to dosing.
* Drug or alcohol addiction requiring treatment in the past 12 months.
* Donation or significant loss of whole blood (480 ml or more) within 30 days or plasma within 14 days prior to dosing.
* Positive test results for HIC, Hepatitis B surface antigen or Hepatitis C antibody.
* Positive test results for drugs of abuse at screening.
* Positive serum pregnancy test.
* Tobacco user within 90 days of the first study dose.
* Unable, or unwilling to tolerate multiple venipunctures.
* Difficulty fasting or eating the standard meals that will be provided.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2004-11; Primary Completion 2004-11 (Actual); Study Completion 2004-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: So Ran Hong, M.D., Principal Investigator — Novum Pharmaceutical Research Services
Locations (1):
- Novum Pharmaceutical Research Services, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Test (Ropinirole HCl) First: 0.25 mg Ropinirole HCl Tablets test product dosed in first period followed by 0.25 mg Requip® Tablets reference product dosed in the second period.
- Reference (Requip®) First: 0.25 mg Requip® Tablets reference product dosed in first period followed by 0.25 mg Ropinirole HCl Tablets test product dosed in the second period.
Period: First Intervention
Arm/Group | Test (Ropinirole HCl) First | Reference (Requip®) First
Started | 23 | 23
Completed | 23 | 23
Not Completed | 0 | 0
Period: Washout of 7 Days
Arm/Group | Test (Ropinirole HCl) First | Reference (Requip®) First
Started | 23 | 23
Completed | 22 | 22
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1
Period: Second Intervention
Arm/Group | Test (Ropinirole HCl) First | Reference (Requip®) First
Started | 22 | 22
Completed | 22 | 22
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Test (Ropinirole HCl) First | Reference (Requip®) First | Total
Number analyzed (Participants) | 23 | 23 | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 23 | 23 | 46
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 11 | 21
  Male | 13 | 12 | 25
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 1 | 0 | 1
  Black | 13 | 16 | 29
  White | 4 | 2 | 6
  Hispanic | 5 | 5 | 10
Region of Enrollment [Number; unit: participants]
  United States | 23 | 23 | 46

OUTCOME MEASURES:

1. Primary Outcome: Cmax (Maximum Observed Concentration of Drug Substance in Plasma)
Description: Bioequivalence based on Cmax.
Time Frame: Blood samples collected over a 24 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: pg/mL
Groups:
- Test (Ropinirole HCl): 0.25 mg Ropinirole HCl Tablets test product dosed in either period.
- Reference (Requip®): 0.25 mg Requip® Tablets reference product dosed in either period.
Arm/Group | Test (Ropinirole HCl) | Reference (Requip®)
Number analyzed (Participants) | 44 | 44
pg/mL | 564.09 (174.53) | 543.71 (168.9)
Statistical Analysis 1: Comparison: Test (Ropinirole HCl) vs Reference (Requip®); Test type: Non-Inferiority or Equivalence — The ANOVA model was utilized in comparing the effects between the test and reference products. Differences were declared statistically significant at the 5% level (p<0.05); Ratio of the T/R geometric mean x 100 = 103.53, 90% CI [99.16 to 108.09] — Bioequivalence is established if the 90% confidence interval for the ln-transformed geometric mean between the reference and test product fall within the interval of 80-125%

2. Primary Outcome: AUC0-t (Area Under the Concentration-time Curve From Time Zero to Time of Last Measurable Concentration)
Description: Bioequivalence based on AUC0-t.
Time Frame: Blood samples collected over a 24 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: pg*h/mL
Arm/Group | Test (Ropinirole HCl) | Reference (Requip®)
Number analyzed (Participants) | 44 | 44
pg*h/mL | 4300.07 (1960.43) | 4209.47 (1929.76)
Statistical Analysis 1: Comparison: Test (Ropinirole HCl) vs Reference (Requip®); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of the T/R geometric mean x 100 = 102.3, 90% CI [97.56 to 107.27] — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: AUC0-inf (Area Under the Concentration-time Curve From Time Zero to Infinity)
Description: Bioequivalence based on AUC0-inf.
Time Frame: Blood samples collected over a 24 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: pg*h/mL
Arm/Group | Test (Ropinirole HCl) | Reference (Requip®)
Number analyzed (Participants) | 44 | 44
pg*h/mL | 4551.89 (2198.95) | 4441.31 (2139.77)
Statistical Analysis 1: Comparison: Test (Ropinirole HCl) vs Reference (Requip®); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of the T/R geometric mean x 100 = 102.54, 90% CI [97.53 to 107.8] — [estimate comment as in outcome 1, analysis 1]

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Principal Investigator is not permitted to discuss or publish trial results.